CLINICAL TRIAL: NCT00811512
Title: Fundus Changes in the Microphthalmy Eyes
Status: Completed | Type: Observational
Sponsor: Hospital de Olhos Sadalla Amin Ghanem (Other)
Responsible Party: Fernando Jose De Novelli, Fernando Jose De Novelli
Other Study IDs: sadalla1
Record Dates: First submitted 2008-12-18; First posted 2008-12-19 (Estimated); Last update posted 2008-12-19 (Estimated); Status verified 2008-12

CONDITIONS: Eye Diseases, Hereditary
Keywords: retina; fold; fovea
MeSH Terms: conditions — Eye Diseases, Hereditary

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The goal is to describe the fundamental aspects of fundoscopic eye in patients with microphthalmia

DETAILED DESCRIPTION:
Microphthalmos is a developmental ocular disorder defined as a small eyeball. The condition can be associated with abnormalities of anterior and posterior segments. The most common anterior characteristics include corneal opacities, angle-closure and a shallow anterior chamber and cataract. The main findings of posterior segment are uveal effusion, retinal folds, abnormalities of macular capillary vascularization, absence of foveal depression and peripheral retinoschisis. We performed on 3 patients with microphthalmos and their OCT features of posterior segment.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of microphthalmia

Exclusion Criteria:

* Eyes larger than 18mm

Ages: 10 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: the study is the description of three cases of microphthalmy with changes to fund of the eye, all documented with optical coherence tomography and clinical characteristics.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2007-05; Primary Completion 2008-09 (Actual); Study Completion 2008-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Fernando J Novelli, Bsc, Principal Investigator — Hospital de Olhos Sadalla Amin Ghanem